CLINICAL TRIAL: NCT02651064
Title: USDA Healthy Incentives Pilot (HIP)
Brief Title: USDA Healthy Incentives Pilot
Acronym: HIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abt Associates (Industry)
Collaborators: Tufts University (Other); MAXIMUS (Unknown); USDA Food and Nutrition Service (U.S. Federal Agency); Massachusetts Department of Transitional Assistance (Other)
Responsible Party: Principal Investigator, Susan Bartlett, Principal Associate, Abt Associates
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HIP
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Dietary Modification
Keywords: Supplemental Nutrition Assistance Program (SNAP); fruits and vegetables; price incentive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIP (Experimental): Received a 30% rebate on targeted fruits and vegetables (TFV) purchased using SNAP benefits in participating retailers. TFV earning the rebate included fresh, canned, frozen, and dried fruits and vegetables without added sugars, fats, oils, or salt, excluding white potatoes, mature legumes (dried beans and peas), and 100% juice.
  Interventions: Other: HIP
- Non-HIP (No Intervention): Received SNAP benefits as usual.

INTERVENTIONS:
Other: HIP
  Other Names: Healthy Incentives Pilot; Financial incentives; Rebate; Price intervention
  Arms: HIP

SUMMARY:
The USDA Healthy Incentives Pilot (HIP) evaluated the impact of a 30% financial incentive on fruit and vegetable intake among adult participants in the USDA Supplemental Nutrition and Assistance Program (SNAP).

DETAILED DESCRIPTION:
U.S. fruit and vegetable intake remains below recommendations, particularly for low-income populations. Evidence on effectiveness of financial incentives for addressing this shortfall is limited.

This study examined effects of USDA's Healthy Incentives Pilot (HIP), which offered financial incentives to Supplemental Nutrition Assistance Program (SNAP) participants for purchasing targeted fruits and vegetables (TFV).

A randomized controlled trial of HIP was conducted in Hampden County, Massachusetts. 7,500 randomly selected SNAP households received a 30% rebate on TFV purchased using SNAP benefits. The remaining 47,595 SNAP households in the county received benefits as usual. Adults in 5,076 households were randomly sampled to complete telephone surveys, including 24-h dietary recall interviews. Surveys were conducted at baseline-1-3 mo pre-implementation-and in two follow-up rounds, 4-6 mo and 9-11 mo post-implementation. 2,784 adults (1,388 HIP, 1,396 non-HIP) completed baseline interviews; data were analyzed for 2,009 adults (72%) also completing at least one follow-up interview.

ELIGIBILITY:
Inclusion Criteria:

* Households with residential or mailing address in Hampden County, Massachusetts
* Receiving SNAP benefits in July 2011

Exclusion Criteria:

* Child-only cases (households not including at least one member aged 16 or older eligible to serve as SNAP head of household)
* Cases with benefits signed over to residential or treatment facilities

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55095 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Targeted fruit and vegetable (TFV) intake | Intake in prior 24 hours; assessed in two follow-up rounds (4-6 mo and 9-11 mo post-implementation) with 10% replicate subsample in each round; data pooled across two follow-up rounds and replicate samples for primary analysis
  Daily adult intake of fresh, canned, frozen, and dried fruits and vegetables without added sugars, fats, oils, or salt, excluding white potatoes, mature legumes (dried beans and peas), and 100% juice.
  In total and by USDA food pattern group (all targeted fruits; citrus, melon, and berries; other fruits; all targeted vegetables; dark green vegetables; red & orange vegetables (including tomatoes and other red & orange vegetables); starchy vegetables (excluding white potatoes); and other vegetables.)
  Assessed via computer-assisted telephone interview 24-hour dietary recall (Automated Multiple Pass Method).
  Measured in cup-equivalents based on USDA Food Pattern Equivalents Database (FPED).
  Secondary analyses assessed changes between follow-up rounds.

SECONDARY OUTCOMES:
All fruit and vegetable intake | Intake in prior 24 hours; assessed in two follow-up rounds (4-6 mo and 9-11 mo post-implementation) with 10% replicate subsample in each round; data pooled across two follow-up rounds and replicate samples for main analysis
  Daily adult intake of all fruits and vegetables (fresh, canned, frozen, or dried).
  In total and by USDA food pattern group (all fruits; citrus, melon, and berries; other fruits; all vegetables; dark green vegetables; red & orange vegetables (including tomatoes and other red & orange vegetables); starchy vegetables (including white potatoes and other starchy vegetables); legumes; and other vegetables.)
  Assessed via computer-assisted telephone interview 24-hour dietary recall (Automated Multiple Pass Method).
  Measured in cup-equivalents based on USDA Food Pattern Equivalents Database (FPED).
  Secondary analyses assessed changes between follow-up rounds.
Intake of other foods | Intake in prior 24 hours; assessed in two follow-up rounds (4-6 mo and 9-11 mo post-implementation) with 10% replicate subsample in each round; data pooled across two follow-up rounds and replicate samples for main analysis
  Daily adult intake of other foods.
  By USDA food pattern group (total grains (including whole and refined grains) (ounce-equivalents); total dairy (cup-equivalents); total protein foods (ounce-equivalents); total oils (gram-equivalents); solid fats (gram-equivalents); added sugars (teaspoons); and alcoholic drinks (drinks)).
  Assessed via computer-assisted telephone interview 24-hour dietary recall (Automated Multiple Pass Method).
  Measured in servings based on units as specified in the USDA Food Pattern Equivalents Database (FPED).
  Secondary analyses assessed changes between follow-up rounds.
HEI-2010 | Calculated based on intake in prior 24 hours; assessed in two follow-up rounds (4-6 mo and 9-11 mo post-implementation) with 10% replicate subsample in each round; data pooled across two follow-up rounds and replicate samples for main analysis
  Healthy Eating Index-2010 (Guenther et al. 2014).
  Total and component scores (total fruit; whole fruit; total vegetables; beans and greens; whole grains; dairy; total protein foods; seafood and plant proteins; fatty acids; refined grains; sodium; empty calories).
  Assessed via computer-assisted telephone interview 24-hour dietary recall (Automated Multiple Pass Method).
  Servings calculated based on units as specified in the USDA Food Pattern Equivalents Database (FPED).
  Estimated via population ratio method (see Freedman et al. 2010).
  Secondary analyses assessed changes between follow-up rounds.

OTHER OUTCOMES:
Family food environment | Assessed at baseline (1-3 mo prior to implementation) and two follow up rounds (4-6 mo and 9-11 mo post-implementation); data pooled across two follow-up rounds for main analysis
  Series of nine individual categorical measures describing current family food environment.
  Assessed via computer-assisted telephone interview.
  Survey items:
  "How often do you...
  * Have fruit available at home?
  * Have fruit in refrigerator or on counter?
  * Have vegetables available at home?
  * Have ready-to-eat vegetables in fridge or on counter?
  * Have salty snacks at home (chips, crackers)?
  * Have lowfat/nonfat milk at home?
  * Have soft drinks/fruit drinks (not juice) at home?
  * Sit down with family at home for evening meals?
  * Cook evening meals at home?"
  Response categories: 1=never/no refrigerator or freezer, 2=rarely, 3=sometimes, 4=most of the time, 5=always.
  Secondary analyses assessed changes between follow-up rounds. Baseline values used as covariates in impact estimation regression models to improve precision.
Exposure to nutrition education and promotion | Past 3 months; assessed at baseline (1-3 mo prior to implementation) and two follow up rounds (4-6 mo and 9-11 mo post-implementation); data pooled across two follow-up rounds for main analysis
  Two individual binary measures describing exposure to nutrition education and promotion in prior three months.
  Assessed via computer-assisted telephone interview.
  Survey items:
  "In the past three months, have you...
  * heard or seen messages about fruits & vegetables?
  * attended a nutrition education class or program?"
  Response categories: 1=yes, 2=no.
  Secondary analyses assessed changes between follow-up rounds. Baseline values used as covariates in impact estimation regression models to improve precision.
Food preferences and beliefs | Assessed at baseline (1-3 mo prior to implementation) and two follow up rounds (4-6 mo and 9-11 mo post-implementation); data pooled across two follow-up rounds for main analysis
  Six individual 5-point Likert scales describing current food preferences and beliefs.
  Assessed via computer-assisted telephone interview.
  Survey items:
  "How much do you agree or disagree with the following statements?
  * I enjoy trying new foods.
  * I enjoy trying new fruits.
  * I enjoy trying new vegetables.
  * I eat enough fruits to keep me healthy.
  * I eat enough vegetables to keep me healthy.
  * I often encourage family/friends to eat fruits & vegetables."
  Response categories: 1=strongly disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, 5=strongly agree.
  Secondary analyses assessed changes between follow-up rounds. Baseline values used as covariates in impact estimation regression models to improve precision.
Perceived barriers to fruit and vegetable consumption | Assessed at baseline (1-3 mo prior to implementation) and two follow up rounds (4-6 mo and 9-11 mo post-implementation); data pooled across two follow-up rounds for main analysis
  Seven individual 5-pt Likert scales re: barriers to fruit & vegetable consumption.
  Assessed via computer-assisted telephone interview.
  Svy items:
  "How much do you agree/disagree that
  * It's hard to eat vegetables b/c I don't know how to prepare them.
  * It's hard to eat vegetables b/c they are hard to find where I shop.
  * It's hard to eat fruits b/c they are hard to find where I shop.
  * I don't eat fruits & vegetables as much as I would like b/c they cost too much.
  * I don't eat fruits & vegetables as much as I would like b/c they spoil.
  * I don't eat fruits & vegetables as much as I would like b/c my family dislikes them.
  * I don't eat fruits & vegetables as much as I would like b/c I don't like them."
  Responses: 1=strongly disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, 5=strongly agree.
  Secondary analyses assessed changes btw follow-up rounds. Baseline values used as covariates in impact regression models to improve precision.
Perceived barriers to grocery shopping | Assessed at baseline (1-3 mo prior to implementation) and two follow up rounds (4-6 mo and 9-11 mo post-implementation); data pooled across two follow-up rounds for main analysis
  Two individual 5-point Likert scales describing perceived barriers to grocery shopping.
  Assessed via computer-assisted telephone interview.
  Survey items:
  "How often are you kept from grocery shopping by...
  * limited transportation?
  * the distance to the grocery store?"
  Response categories: 1=never, 2=rarely, 3=sometimes, 4=most of the time, 5=always.
  Secondary analyses assessed changes between follow-up rounds. Baseline values used as covariates in impact estimation regression models to improve precision.
Average monthly household Supplemental Nutrition Assistance Program (SNAP) food expenditures | Assessed for two follow up rounds (4-6 mo and 9-11 mo post-implementation); data pooled across two follow-up rounds for main analysis
  Constructed from SNAP electronic benefit transfer (EBT) transactions data for March-October 2012.
  * Household SNAP expenditures per month (total, by retailer type: supermarkets/ superstores, convenience, grocery, farmers markets, other, out of state; and by HIP participation (HIP participating retailers and nonparticipating retailers)
  * Household SNAP expenditures per month on targeted fruits and vegetables, including fresh, canned, frozen, and dried fruits and vegetables without added sugars, fats, oils, or salt, excluding white potatoes, mature legumes (dried beans and peas), and 100% juice.
  Secondary analyses assessed changes between follow-up rounds.
Self-reported monthly household expenditures | Assessed at baseline (1-3 mo prior to implementation) and two follow up rounds (4-6 mo and 9-11 mo post-implementation); data pooled across two follow-up rounds for main analysis
  Self-reported monthly household expenditures, by category.
  Assessed via computer-assisted telephone interview.
  Survey item:
  "Please tell us how much you usually spend per month on....
  * Groceries using only SNAP
  * Groceries not using SNAP
  * Nonfood items
  * Restaurants
  * All fruits and vegetables"
  Secondary analyses assessed changes between follow-up rounds. Baseline values used as covariates in impact estimation regression models to improve precision.
Usual grocery shopping location | Assessed at baseline (1-3 mo prior to implementation) and two follow up rounds (4-6 mo and 9-11 mo post-implementation); data pooled across two follow-up rounds for main analysis
  Usual store type for grocery shopping.
  Assessed via computer-assisted telephone interview.
  Survey item:
  "Where do you usually go grocery shopping?
  * Large chain grocery store or supermarket
  * Discount superstore (such as Walmart)
  * Small local store or corner store
  * Warehouse club store (such as Sam's Club or Costco)
  * Natural or organic supermarket (such as Whole Foods Market)
  * Ethnic market
  * Farmers market/co-op
  * Convenience store (such as 7-11 or mini market)
  * Some other location (specify)."
  Secondary analyses assessed changes between follow-up rounds. Baseline values used as covariates in impact estimation regression models to improve precision.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bartlett, PhD, Principal Investigator — Abt Associates

IPD SHARING:
Plan to Share IPD: Yes
Public use dataset available by request from USDA Food & Nutrition Service.

REFERENCES:
- [Background] Abt Associates Inc. Healthy Incentives Pilot: Updated Study Plan. USDA, Food and Nutrition Service, 2011. http://www.fns.usda.gov/sites/default/files/study_plan.pdf.
- [Background] Bartlett S, Beauregard M, Logan C, Komarovsky M, Wommack T, Wilde P, Owens C, Melham M, McLaughlin T. Healthy Incentives Pilot (HIP): Early Implementation Report. USDA, Food and Nutrition Service, 2013. http://www.fns.usda.gov/sites/default/files/HIP_Early_Implementation.pdf.
- [Background] Chu, A. Evaluation of the Healthy Incentives Pilot (HIP): Participant survey weighting methodology. Alexandria, VA: USDA, Food and Nutrition Service, Office of Policy Support, 2014.
- [Result] Bartlett S, Klerman J, Olsho L, Logan C, Blocklin M, Beauregard M, Enver A, Wilde P, Owens C, Melhem M. Evaluation of the Healthy Incentives Pilot (HIP): Final Report. USDA, Food and Nutrition Service, 2014. http://www.fns.usda.gov/healthy-incentives-pilot-final-evaluation-report.
- [Result] Wilde P, Klerman JA, Olsho LEW, Bartlett S. Explaining the impact of USDA's Healthy Incentives Pilot on different spending outcomes. Appl Econ Perspect Policy 2015 (Epub ahead of print; DOI: Epub ahead of print; DOI: doi:10.1093/aepp/ppv028).
- [Result] Klerman JAK, Bartlett S, Wilde P, Olsho L. The short-run impact of the Healthy Incentives Pilot Program on fruit and vegetable intake. Am J Agr Econ 2015;96:1372-82.
- [Derived] Olsho LE, Klerman JA, Wilde PE, Bartlett S. Financial incentives increase fruit and vegetable intake among Supplemental Nutrition Assistance Program participants: a randomized controlled trial of the USDA Healthy Incentives Pilot. Am J Clin Nutr. 2016 Aug;104(2):423-35. doi: 10.3945/ajcn.115.129320. Epub 2016 Jun 22. PMID 27334234